CLINICAL TRIAL: NCT04804579
Title: Boston Alcohol Research Collaboration on HIV/AIDS (ARCH) Frailty, Functional Impairment, Falls, and Fractures (4F) Fall Prevention Intervention Pilot Study
Brief Title: Boston ARCH 4F Intervention to Reduce Fall Risk in People With HIV and Alcohol Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-41041; U01AA020784 (NIH)
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: HIV Infection; Alcohol Consumption; Falls, Accidental; Falls
Keywords: HIV Infection; Alcohol Consumption; Falls, Accidental; Falls; Substance Use; Intervention Study
MeSH Terms: conditions — HIV Infections; Alcohol Drinking; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fall Prevention Intervention (Experimental): The Intervention involves 3 primary components: virtual group sessions, at-home exercises, and weekly phone check-ins.
  Virtual Group Session will be held via phone/video call for approximately 30 minutes per week for 10 weeks.
  At-Home Exercises will be assigned by a registered occupational therapist member of the study team, and participants will be instructed to complete them independently at home 3 times per week. Participants will record the exercises that they complete.
  Weekly Phone Check-Ins will occur once per week. These check-ins will be used to provide support and problem solving as needed, and individualized reminder systems will be set up to prompt the participant to engage in their weekly exercises (e.g., set up alarm on phone, notifications through calendar app).
  Interventions: Behavioral: Fall Prevention Intervention
- Control Group (No Intervention): Participants will be provided with an educational pamphlet that includes resources related to falls and alcohol use.

INTERVENTIONS:
Behavioral: Fall Prevention Intervention — The intervention will aim to reduce fall risk through weekly virtual group meetings and at-home exercise assignments to address physical and environmental factors that may put participants at a higher risk of experiencing a fall.
  Arms: Fall Prevention Intervention

SUMMARY:
This study is being conducted to assess the acceptability and feasibility of a randomized trial of a 10 week virtual intervention to reduce fall risk in people with HIV who consume alcohol. The hypothesis is that this randomized trial of the fall prevention intervention will be found to be feasible and acceptable in this pilot stage.

Standardized assessments will be administered in-person at Boston University Medical Campus to assess various domains including fall risk, fear of falling, physical performance measures (such as grip strength, balance, and gait speed), substance use, and other related measures. The intervention has 3 main components: home exercises, virtual group sessions and weekly phone check-ins. Home exercise will be customized to match the current fitness level of participants. Participants will be asked to complete assigned exercises 3 times per week. Additionally, there will be a weekly virtual group session led by an Occupational Therapist trained in group facilitation via Zoom. The virtual group sessions will be used to help answer any questions and lead a discussion around challenges related to falls. Finally, a member of the research team will check-in with participants once per week to answer any remaining questions that participants have, provide individual feedback on exercises, and set up reminders for the upcoming week. Reminders will be tailored to the individual participant's needs to remind the participant to complete the intervention's components.

ELIGIBILITY:
Inclusion Criteria:

* Prior or current participant in the Boston ARCH 4F Cohort
* Any alcohol consumption in the last 30 days using Addiction Severity Index
* Deemed a Fall Risk using the CDC STEADI Fall Risk Assessment Form
* Has reliable access to a phone or computer with internet connection

Exclusion Criteria:

* Requires wheelchair for mobility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa W Kim, MD, Principal Investigator — Boston University; Simone Gill, PhD, Study Director — Boston University
Locations (1):
- Boston University Medical Campus, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gill SV, Shin D, Kim TW, Magane KM, Hereen T, Winter M, Helfrich C, Saitz R. A Fall Prevention Feasibility Trial for People With HIV and Alcohol Use. OTJR (Thorofare N J). 2025 Jan;45(1):85-94. doi: 10.1177/15394492241238956. Epub 2024 Mar 30. PMID 38554013
- [Derived] Shin D, Gill SV, Kim TW, Magane KM, Mason T, Heeren T, Winter M, Helfrich C, Saitz R. Study Protocol for a Pilot Randomized Trial of a Virtual Occupational Therapy Fall Prevention Intervention for People With HIV and Alcohol Use. Subst Abuse. 2022 Dec 23;16:11782218221145548. doi: 10.1177/11782218221145548. eCollection 2022. PMID 36578450

RESULTS

PARTICIPANT FLOW:
Groups:
- Fall Prevention Intervention: The Intervention involves 3 primary components: virtual group sessions, at-home exercises, and weekly phone check-ins.
  Virtual Group Session will be held via phone/video call for approximately 30 minutes per week for 10 weeks.
  At-Home Exercises will be assigned by a registered occupational therapist member of the study team, and participants will be instructed to complete them independently at home 3 times per week. Participants will record the exercises that they complete.
  Weekly Phone Check-Ins will occur once per week. These check-ins will be used to provide support and problem solving as needed, and individualized reminder systems will be set up to prompt the participant to engage in their weekly exercises (e.g., set up alarm on phone, notifications through calendar app).
  Fall Prevention Intervention: The intervention will aim to reduce fall risk through weekly virtual group meetings and at-home exercise assignments to address physical and environmental factors that may put participants at a higher risk of experiencing a fall.
Period: Overall Study
Arm/Group | Fall Prevention Intervention | Control Group
Started | 12 | 11
Completed | 11 | 11
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fall Prevention Intervention | Control Group | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (8.3) | 58.5 (8.2) | 57.9 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Engagement With Intervention
Description: Number of weekly virtual group intervention sessions attended (of 10 sessions)
Time Frame: 10 weeks (final assessment)
Population: Analysis population includes participants assigned to the Fall Prevention Intervention who completed the 10-week follow-up research assessment.
Measure: Mean (Standard Deviation); unit: intervention sessions
Arm/Group | Fall Prevention Intervention | Control Group
Number analyzed (Participants) | 11 | 0
intervention sessions | 3.27 (3.44) |

2. Primary Outcome: Satisfaction With Intervention
Description: Measured using the Client Satisfaction Questionnaire (CSQ-8), which includes 8 items that yield a single score measuring a single dimension of overall satisfaction. Each item is assessed using a Likert scale that ranges from 1-4. Scores range from 8-32, with higher values indicating greater satisfaction.
Time Frame: 10 weeks (final assessment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fall Prevention Intervention | Control Group
Number analyzed (Participants) | 11 | 0
score on a scale | 30.35 (1.57) |

3. Secondary Outcome: Change in Self Reported Falls
Description: A fall is defined as an unexpected event, including a slip or a trip, in which a participant lost their balance and landed on the floor, ground, or lower level, or hit an object like a table or a chair. Participants self-report as having experienced 0 falls, 1 fall, 2 falls, 3-5 falls, or more than 5 falls. Results were dichotomized as no falls, or 1 or more fall. Outcome results are reported as change from baseline to follow-up in the percentage of participants with at least one fall.
Time Frame: Baseline and 10 weeks (final assessment)
Population: Participants who completed the 10-week follow-up research assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Fall Prevention Intervention | Control Group
Number analyzed (Participants) | 11 | 11
Percentage of participants | -38.6 | 0

4. Secondary Outcome: Change in Physical Function Based on the Short Physical Performance Battery Assessment
Description: A composite score based on balance (the ability to stand for 10 seconds with feet in 3 different positions: side-by-side, semi-tandem, and tandem), gait speed (timed trial of a 4m walk), and chair rises (time to rise from a chair 5 times). The score ranges from 0-12, with a higher score indicating better physical function.
Time Frame: Baseline and 10 weeks (final assessment)
Population: Participants who completed the 10-week follow-up research assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fall Prevention Intervention | Control Group
Number analyzed (Participants) | 11 | 11
score on a scale | 0.82 (1.25) | 0.36 (1.29)

5. Secondary Outcome: Change in Fried's Frailty Phenotype
Description: Frailty is defined as the presence of five components: Weakness, defined as having a low grip strength measured with a dynamometer; slowness, defined as having a slow walking speed measured using a 20 meter gait speed assessment; exhaustion, defined as answering "Most or all of the time (5-7 days)" to at least one of two questions from the Center for Epidemiologic Studies (CESD-10) scale ("How often do you feel like everything you did was an effort?" and "How often did you feel like you could not get going?"); Low physical activity, defined as answering "Yes, limited a lot" to the question "Does your health limit you in vigorous activities, such as running, lifting heavy objects, participating in strenuous sports?"; and unintentional weight loss, defined as answering "Yes" to the question "In the past year, have you lost more than 10 pounds unintentionally?". Stages of frailty are categorized as: Non-frail (score 0), Pre-frail (score 1-2), and Frail (score 3-5).
Time Frame: Baseline and 10 weeks (final assessment)
Population: Participants who completed the 10-week follow-up research assessment with complete (non-missing) data on all components of the Frailty Phenotype
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fall Prevention Intervention | Control Group
Number analyzed (Participants) | 11 | 10
score on a scale | -0.09 (1.58) | 0.3 (0.82)

6. Secondary Outcome: Change in Number of Days of Alcohol Use and Other Drug Use in the Past 30 Days
Description: Measured using the past 30 day alcohol/drug use section of the Addiction Severity Index (ASI), a validated instrument. The past 30 day alcohol/drug use section of the ASI measures the number of days of substance use in the past 30 days. The substances assessed by the ASI include: alcohol [number of days where 4+ drinks (women)/5+drinks (men) were consumed], cocaine, heroin, hallucinogens, phencyclidines, cannabis/marijuana, stimulants/amphetamines, tranquilizers/sedatives, non-prescribed buprenorphine, non-prescribed methadone, other non-prescribed prescription opioids, inhalants, synthetic marijuana/K2/spice, miscellaneous. Number of days range from 0-30 for each substance, with a higher number of days indicating more frequent substance use.
Time Frame: Baseline and 10 weeks (final assessment)
Population: Participants who completed the 10-week follow-up research assessment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fall Prevention Intervention | Control Group
Number analyzed (Participants) | 11 | 11
days | -1.36 (5.64) | -0.45 (7.12)

ADVERSE EVENTS:
Time Frame: From enrollment through completion of a participant's 10-week follow-up research assessment window.
Arm/Group | Fall Prevention Intervention | Control Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT04804579/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT04804579/ICF_000.pdf